CLINICAL TRIAL: NCT07369895
Title: A Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Chimeric Antigen Receptor T Cell (O&D-001) Injection Targeting BCMA and GPRC5D in the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Clinical Study of O&D-001 Injection in the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: O&D BioTech Group CO., Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: O&D-001-IIT
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This study presets three dosage groups.Using the traditional 3+3 dose escalation method, 3 - 6 subjects with relapsed or refractory multiple myeloma are planned to be enrolled in each dose group. Dose escalation studies will be conducted sequentially from the low - dose group to the high - dose group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV Dose-Escalation Cohort (Experimental): Single dose administration of O&D-001 via intravenous infusion.
  Interventions: Biological: Chimeric antigen receptor T cell O&D-001 injection targeting BCMA and GPRC5D

INTERVENTIONS:
Biological: Chimeric antigen receptor T cell O&D-001 injection targeting BCMA and GPRC5D — Using the traditional 3+3 dose escalation method.

SUMMARY:
This study is a single-center, open and dose-escalation clinical study to evaluate the safety, tolerability, PK/PD characteristics and preliminary efficacy of the investigational drug O&D-001 injection in the treatment of relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, inclusive, regardless of gender.
2. Subjects voluntarily agree to participate in this study, sign the informed consent form, and are willing to complete all trial procedures.
3. Meets the internationally accepted diagnostic criteria for multiple myeloma (IMWG Diagnostic Criteria 2016, Appendix 1).
4. Tumor specimen (bone marrow) from the subject tests positive for BCMA or GPRC5D expression on the myeloma cell membrane via immunohistochemistry (IHC) or flow cytometry.
5. Patients with multiple myeloma who have received at least 2 prior lines of anti-myeloma therapy, including failure of at least one proteasome inhibitor and one immunomodulatory agent; each line of therapy should have consisted of at least one complete treatment cycle, unless the best response to that therapy was documented as Progressive Disease (PD) (according to the 2016 IMWG Response Criteria, Appendix 1); must have documented PD during or within 12 months after the last line of therapy.
6. Has measurable disease, defined as meeting at least one of the following criteria prior to apheresis: serum M-protein ≥5 g/L; urine M-protein ≥200 mg/24 hours; for subjects with light chain multiple myeloma not meeting the above serum or urine M-protein criteria, an abnormal serum free light chain (sFLC) ratio with involved FLC ≥100 mg/L; >5% clonal plasma cells in bone marrow aspirate or biopsy as assessed by cytology or flow cytometry.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
8. Life expectancy of at least 3 months.
9. Major organ function is normal, defined as meeting the following criteria:

   * Hemoglobin ≥8.0 g/dL (No red blood cell (RBC) transfusion within 7 days prior to laboratory testing; use of recombinant human erythropoietin is allowed. For subjects who meet the inclusion criteria at screening, RBC transfusion is permitted after the first hematology test at screening to maintain hemoglobin level ≥8.0 g/dL.)
   * Platelets ≥50×10⁹/L (No platelet transfusion or transfusion support within 7 days prior to laboratory testing)
   * Absolute Neutrophil Count (ANC) ≥1.0×10⁹/L (Previous use of growth factor support is allowed, but no supportive treatment within 7 days prior to laboratory testing).
   * AST and ALT ≤3.0 × Upper Limit of Normal (ULN).
   * Creatinine Clearance ≥40 mL/min (Cockcroft-Gault formula).
   * Total Bilirubin ≤1.5 × ULN.
   * Corrected Serum Calcium ≤12.5 mg/dL (≤3.1 mmol/L) or Ionized Calcium ≤6.5 mg/dL (≤1.6 mmol/L).
   * Fibrinogen ≥1.0 g/L.
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5×ULN.
   * Prothrombin Time (PT) ≤1.5 × ULN.
   * Oxygen Saturation (on room air, without oxygen supplementation) ≥92%.
   * Left Ventricular Ejection Fraction (LVEF) ≥50%.
10. Subjects with childbearing potential must use at least one medically recognized contraceptive method (e.g., intrauterine device, oral contraceptives, or condoms) during the study treatment period (from screening to 24 months after cell infusion). Female subjects of childbearing age must have a negative serum/urine HCG test within 7 days prior to cell therapy initiation and must not be lactating.

Exclusion Criteria:

1. Prior treatment with CAR-T/TCR-T/TIL or other cell therapies; known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
2. Allergy or intolerance to any of the study drugs (including chemotherapy preconditioning drugs and tocilizumab) or to any component of the cell therapy product.
3. Received systemic anti-tumor therapy within 2 weeks prior to apheresis; or monoclonal antibody therapy for multiple myeloma within 3 weeks prior to apheresis; or radiotherapy within 2 weeks prior to apheresis, unless the radiation field involved ≤5% of the bone marrow reserve, in which case the subject is eligible regardless of the end date of radiotherapy.
4. Participated in another clinical trial within 4 weeks prior to apheresis or within 5 half-lives of the investigational drug (whichever is longer).
5. Use of prednisone >10 mg/day (or equivalent dose of other corticosteroids) within 1 week prior to apheresis.
6. Underwent major surgery within 2 weeks prior to apheresis.
7. Presence of any uncontrolled active infection.
8. Severe cardiac disease, including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] class ≥Ⅲ), or severe arrhythmia.
9. Unstable systemic diseases as judged by the investigator, including but not limited to: uncontrolled hypertension despite medication; severe hepatic, renal, or metabolic diseases requiring pharmacological treatment; autoimmune diseases, immunodeficiency, or other conditions requiring immunosuppressive therapy.
10. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and have a hepatitis B virus (HBV) DNA titer above the lower limit of the normal range of the study center; subjects who are positive for hepatitis C virus (HCV) antibody and have detectable peripheral blood HCV RNA; subjects who are positive for human immunodeficiency virus (HIV) antibody; subjects with positive syphilis testing.
11. Diagnosis of malignancies other than multiple myeloma within 5 years prior to screening (except for carcinoma in situ [e.g., breast, bladder, cervical carcinoma in situ] or basal cell carcinoma or squamous cell carcinoma of the skin that have received potentially curative treatment).
12. Received autologous stem cell transplantation within 12 weeks prior to apheresis.
13. Received live vaccines within 4 weeks prior to apheresis.
14. History of central nervous system (CNS) diseases, such as seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, psychosis; known active or history of CNS involvement or clinical signs indicating meningeal/spinal meningeal involvement by multiple myeloma.
15. Diagnosis of plasma cell leukemia.
16. The investigator deems the subject unsuitable for participation in this clinical study due to any clinical or laboratory abnormality or other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 28 days after the first O&D-001 infusion.
Adverse Events (AE) and Serious Adverse Events (SAE) | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided